CLINICAL TRIAL: NCT05071534
Title: Implementation of the Robson Classification of the Cesearn Section in Sohag University Hospital
Brief Title: Implementation of the Robson Classification of Cesearn Section in Sohag University Hospital
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Sahar Abdelfatah, Principal investigator, Sohag University
Other Study IDs: Soh-Med-21-09-01
Record Dates: First submitted 2021-09-14; First posted 2021-10-08 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2021-10

CONDITIONS: Robson Classification System

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim Of The Work find out the frequency and indications for CS in sohag university hospitals and to analyze them according to Robson' ten group classification. This would be helping in adopting suitable measures to reduce the CS rate and identifying various challenges in our setting.

DETAILED DESCRIPTION:
Cesarean Section Is A Surgical Procedure Used to Deliver A Baby Through Incisions In The Abdomen And Uterus . The incidence of Caesarean deliveries is increasing every day passing faraway beyond WHO recommended rate of 15% for all deliveries(1).

The rates of maternal morbidity and mortality are higher after CS compared to vaginal birth. CS is associated with an increased risk of abnormal placentation, uterine rupture, ectopic pregnancy, stillbirth, and preterm birth.

therefor Increase rate of unnecessary caesarean sections has been a growing concern in most parts of the world,Worldwide Caesarean section rates have risen from around 7% in 1990 to 21% in 2021 and are projected to continue over current decade if this trend continuees,by 2030 the highest rates are likely to be in Eastern Asia(63),Latin America and the Caribbean (54),Western Asia (50), Northen Africa (48),Southern Europe (47) and Australia and New Zealand(45) . According to the latest survey , one in five women in the world now deliver by caesarean section .Egypt has the highest rate of Caesarean section of 54 % in the Eastern Mediterranean Region , with no furthermore improvement to maternal and child mortality rates(2).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women more than 28 wks who will be admitted for labour

Exclusion Criteria:

* pregnant women less than 28wks
* pregnant women presented with rupture uterus

Ages: 15 Years to 45 Years | Sex: Female
Age Groups: Child, Adult
Study Population: Pregnant women more than 28wks who will be admitted for labour in sohag university hospital
Sampling Method: Probability Sample
Enrollment: 1234 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Frequency of cesearn sections in sohag university hospital | Within 6 months
  Number of cesearn sections per year

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag faculty of medicine, Sohag, Egypt